CLINICAL TRIAL: NCT06019884
Title: A Tele-detection and Referral pAthways Model for Early Childhood cariEs Control- a Randomized Factorial Study: The TRACE Study
Brief Title: A Tele-detection and Referral Pathways Model for Early Childhood Caries Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: #1-10/7/2023
Record Dates: First submitted 2023-08-23; First posted 2023-08-31 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Early Childhood Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intraoral camera, conventional referral (Experimental)
  Interventions: Device: Caries detection method: Intraoral camera; Other: Referral pathway: Conventional referral
- Intraoral camera, user fee removal (Experimental)
  Interventions: Device: Caries detection method: Intraoral camera; Other: Referral pathway: User fee removal
- Smartphone camera, conventional referral (Experimental)
  Interventions: Device: Caries detection method: Smartphone camera; Other: Referral pathway: Conventional referral
- Smartphone camera, user fee removal (Experimental)
  Interventions: Device: Caries detection method: Smartphone camera; Other: Referral pathway: User fee removal

INTERVENTIONS:
Device: Caries detection method: Intraoral camera — A specialized intraoral camera (C50) with fluorescence signal and selective chromatic amplification will be used to record intraoral structures in the form of videos and/or photos. The camera has four modes (Daylight, Daylight+, Perio and Caries modes) which can differentiate the color of tissues to provide a reliable diagnosis. The camera will be used in a systemic sequence to video record and capture photos of intraoral conditions in both arches. The intraoral camera will be connected to a laptop screen, and the captured videos and/ or photos will be transferred to an electronic platform.
  Arms: Intraoral camera, conventional referral; Intraoral camera, user fee removal
Device: Caries detection method: Smartphone camera — This is a low-cost electronic system consisting of a smartphone positioned in front of the oral cavity to scan the upper and lower jaws from the cheek then the tongue sides. The smartphone camera resolution should be sensitive enough to capture the intraoral structures (at least 1000 pixels). The focus will be adjusted, and the inbuilt flash will be used to obtain clear and sharp images. The photos will be transferred to the electronic platform.
  Arms: Smartphone camera, conventional referral; Smartphone camera, user fee removal
Other: Referral pathway: User fee removal — The child's parent/ legal guardian will receive financial incentives. These a are designed to cover the costs of treatment and transportation and are tied to attending the preventive dental visit. The child will receive complete dental care.
  Arms: Intraoral camera, user fee removal; Smartphone camera, user fee removal
Other: Referral pathway: Conventional referral — Children will be referred without providing financial incentives following the current standard of care in dental clinics in the public sector in Egypt. Care is planned by the receiving/ treating dentist, based on available resources, and hospital/ clinic policies. The screening/ sending dentist will inform the family about the oral health condition/s and planned treatment costs for which the child needs care and of available public and private facilities that offer the required care.
  Arms: Intraoral camera, conventional referral; Smartphone camera, conventional referral

SUMMARY:
The aim of the study is to assess the effectiveness of ECC tele-detection methods combined with referral pathways, with and without user fee removal, in controlling ECC.

ELIGIBILITY:
Inclusion Criteria:

* Age <6 years old with primary dentition only.
* Written consent from the legal guardian

Exclusion Criteria:

* Children above 6 years old.
* Children with mixed or permanent dentitions.
* Children with physical disabilities or psychiatric disorders.
* Children with intellectual disabilities.
* Children indicated for dental treatment under general anesthesia

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of teeth receiving care | up to 12 months
  This will be assessed using the Caries Assessment Spectrum and Treatment (CAST) index. The CAST index hierarchically describes the full spectrum of caries from the absence of caries, passing through prevention (sealants) and treatment (restoration), to the presence of carious lesions with their complications (pulp exposure, abscess/fistula, and tooth loss). As for the condition severity, Codes 0-2 represent "healthy", 3 indicates "pre-morbidity", while 4-5 indicate "morbidity", 6-7 indicate "serious morbidity", and 8 indicates "mortality".

SECONDARY OUTCOMES:
Oral health-related quality of life | up to 12 months
  This will be assessedusing the Arabic Version of Early Childhood Oral Health Impact Scale (ECOHIS).The scale comprises 13 items included in two main sections: the Child Impact Section (9 items) and the Family Impact Section (4 items). The Child Impact Section has four domains: child symptom (one item), child function (four items), child psychology (two items) and child self-image and social interaction (two items). The Family Impact Scale has two domains: Parental distress (two items) and Family function (two items). The response options are coded: 0 = never; 1 = hardly ever; 2 = occasionally; 3 = often; 4 = very often. ECOHIS scores are calculated by summing the response codes for the child and family sections separately. The values range from 0 to 52 for the total scale (0-36 for the child section and 0-16 for the family section). The highest score expressed a greater impact of the state of oral health indicating worse quality of life.
Procedure time | throughout the procedure completion
  The time needed for intra-oral scanning and assessing the CAST codes will be recorded per patient, and the average time will be calculated and compared between the two methods.
The child's behavior during dental photography | throughout the procedure completion
  This will be assessed through direct observation of the patients and will be assessed on a 5-point Likert scale ranging from "not at all" to "extremely". Higher scores on the positive items indicate favorable behavior
The child's mood during dental photography | throughout the procedure completion
  This will be assessed based on the modified "Positive and Negative Affect Schedule" (PANAS) scale through direct observation of the patients and will be assessed on a 5-point Likert scale ranging from "not at all" to "extremely". Higher scores on the positive outcomes indicate a better mood, while lower scores on the negative items indicate a worse mood.
Percentage of preventive visits completed per child | up to 12 months
  The number of preventive visits that are attended per child will be assessed.
Rate of treatment completion | up to 12 months
  Treatment completion rate will be assessed by monitoring the procedures received out of all procedures the child was indicated to receive.

CONTACTS AND LOCATIONS:
Overall Officials: Nourhan M Aly, M.Sc, Principal Investigator — Alexandria University; Mona K El Kashlan, PhD, Study Chair — Alexandria University; Nicolas Giraudeau, Study Chair — University Hospital Center of Montpellier, France; Maha El Tantawi, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Aly NM, El Kashlan MK, Giraudeau N, El Tantawi M. Children's Acceptance of Intraoral Cameras and Smartphones for Caries Detection: A Randomized Controlled Clinical Trial. Int J Paediatr Dent. 2025 Jul;35(4):792-799. doi: 10.1111/ipd.13291. Epub 2024 Dec 31. PMID 39737579
- [Derived] Aly NM, El Kashlan MK, Giraudeau N, El Tantawi M. A Tele-detection and referral pAthways model for early childhood cariEs control- a protocol for a randomized factorial study: the TRACE study. BMC Oral Health. 2024 Aug 11;24(1):934. doi: 10.1186/s12903-024-04706-8. PMID 39129017